CLINICAL TRIAL: NCT00668499
Title: A Phase I/II Study of VEGF-Antisense Oligonucleotide (VEGF-AS, Veglin) in Combination With Pemetrexed and Cisplatin for the Treatment of Advanced Malignant Mesothelioma
Brief Title: A Study of VEGF-Antisense Oligonucleotide in Combination With Pemetrexed and Cisplatin for the Treatment of Advanced Malignant Mesothelioma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: University of Southern California (Other)
Collaborators: Sponsor Name Pending (Industry)
Responsible Party: Dr. Barbara Gitlitz, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18M-07-2
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: VEGF-Antisense Oligonucleotide , Pemetrexed, Cisplatin — VEGF-AS either 100 or 200mg/m2 IV days 1-5, Pemetrexed 500mg/m2 and Cisplatin 75mg/m2 IV on day 1. Cycle repeated every 3 weeks until 6 cycles completed, unless PD or toxicities

SUMMARY:
This will be a single institution non-randomized phase I/II trial for patients with malignant mesothelioma stage II and above, who have not received prior chemotherapy for their disease.

The purpose of this phase is to select a dose of VEGF-AS (antiangiogenesis drug)to be given with standard doses of pemetrexed followed by cisplatin on day 1 of a 21-day cycle.

DETAILED DESCRIPTION:
The Study Objectives in Phase I are:

To determine the safety of the combination of VEGF-Antisense Oligonucleotide (VEGF-AS, Veglin™) plus Pemetrexed and Cisplatin in subjects with advanced Malignant Mesothelioma,.via a dose escalation protocol. To determine the Maximum Tolerated Dose (MTD) and Dose Limiting Toxicity (DLT) of VEGF-AS plus Premetrexed and Cisplatin. To determine the time to disease progression To determine the objective response rate of the combination of VEGF-AS plus Pemetrexed and Cisplatin for the treatment of advanced malignant mesothelioma

The study Objectives in Phase II are:

To further characterize the toxicity experienced by patients with malignant mesothelioma treated with VEGF-AS plus Cisplatin and Pemetrexed.

To determine median and overall survival.

The Laboratory objectives are:

To measure plasma VEGF levels before, during, and after therapy as a correlate of outcome. To determine the pharmacokinetic profile of VEGF-AS plus Pemetrexed and Cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant pleural mesothelioma, epithelial, sarcomatoid, or mixed subtype
* Patients must have measurable disease,using RECIST criteria.Pleural effusions and ascites are not considered measurable lesions.
* Patients with pleural mesothelioma must be IMIG stage ≥II
* Age greater than or equal to 18 years.
* ECOG performance status less than or equal to 2 and an estimated survival of at least 3 months
* Patients must have adequate organ and marrow function as defined below:

Absolute neutrophil count greater than or equal to1,500 Platelets greater than or equal to 100,000 Total bilirubin less than or equal to2.0x the upper limits of institutional normal AST/ALT less than or equal to 2.0x the upper limits of institutional normal Creatinine Clearance greater than 50ml/min

* The effects of VEGF-AS on the developing human fetus are unknown.
* Pemetrexed may cause fetal harm when administered to a pregnant woman and is classified pregnancy category D. There are no studies of pemetrexed in pregnant women. Cisplatin is also categorized as FDA Pregnancy Category D. There is positive evidence of human fetal risk. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.
* Patients with history of prior cured malignancy > 5 years since the completion of treatment may be accrued provided that other eligibility criteria are met.

Exclusion Criteria:

* Patients who have had chemotherapy for Mesothelioma prior to study entry
* Patients who have had radiation therapy within 3 weeks prior to entering the study. All patients should have recovered from all toxicities of prior therapy.
* Patients receiving therapy with other investigational agents at the time of study enrollment.
* Patients with uncontrolled brain metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and nursing women are excluded from this study
* Patients who had any major surgery within 4 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the phase II trial will be time to progression | Tumor measurements every 6 weeks

SECONDARY OUTCOMES:
Secondary endpoints are objective response rate and overall survival | Every 6 weeks evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gitlitz, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States